CLINICAL TRIAL: NCT03110900
Title: A Randomized Double-blind Multicenter Double-dummy Non-inferiority Trial of Inhaled Loxapine and Intramuscular Haloperidol + Lorazepam for the Reduction of Agitation
Brief Title: Inhaled Loxapine vs Intramuscular (IM) Haloperidol + Lorazepam for Agitation
Acronym: loxapine
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor Withdrawal
Sponsor: University of Arkansas (Other)
Collaborators: Mount Sinai Hospital, Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 206292
Record Dates: First submitted 2017-03-16; First posted 2017-04-12 (Actual); Results first posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-05

CONDITIONS: Agitation,Psychomotor; Haloperidol Causing Adverse Effects in Therapeutic Use; Lorazepam Causing Adverse Effects in Therapeutic Use; Loxapine Causing Adverse Effects in Therapeutic Use
MeSH Terms: conditions — Psychomotor Agitation | interventions — Haloperidol; Lorazepam; Loxapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- haloperidol + lorazepam (Active Comparator): IM haloperidol 5mg + IM lorazepam 2mg + placebo inhaler
  Interventions: Drug: Haloperidol + lorazepam
- loxapine (Experimental): Inhaled loxapine 10mg + IM normal saline
  Interventions: Drug: Loxapine

INTERVENTIONS:
Drug: Haloperidol + lorazepam — Haloperidol + lorazepam + placebo
  Other Names: Haldol + Ativan
  Arms: haloperidol + lorazepam
Drug: Loxapine — loxapine + placebo
  Other Names: Adasuve
  Arms: loxapine

SUMMARY:
The primary objective of this study is to determine the noninferiority of inhaled loxapine compared to intramuscular haloperidol/lorazepam on agitation reduction at 120 minutes.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the noninferiority of inhaled loxapine compared to intramuscular haloperidol/lorazepam on agitation reduction at 120 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Requires treatment for agitation in the judgment of a physician
2. Patient either pre-consented, has surrogate consent, or able to consent (in cases of mild agitation).
3. The patient is at least 18 years of age and less than 65 years of age.
4. Patients with known or presumed schizophrenia or bipolar 1 disorder.

Exclusion Criteria:

1. Patients with acute respiratory signs/symptoms (eg, wheezing).
2. Known diagnosis of Chronic Obstructive Pulmonary Disease (COPD) or asthma or taking meds for asthma or COPD.
3. Female patients who are obviously pregnant or breast-feeding.
4. Medically unstable patients.
5. Patients or surrogates who object to being in the study (even if previously pre-consented).
6. Physician objection to patient enrollment in the study.
7. Prisoners or incarcerated.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Wilson, MD, Principal Investigator — UAMS
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Haloperidol + Lorazepam | Loxapine
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — Sponsor withdrew | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Haloperidol + Lorazepam | Loxapine | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Customized [Count of Participants; unit: Participants]
  >18 years <99 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Reduction of Agitation on Positive and Negative Syndrome Scale (PANSS)
Description: Change in agitation level on the PANSS from baseline up to 120 minutes -- terminated by sponsor before results available
Time Frame: 120 minutes
Population: No data was collected because the sponsor terminated the study before any data could be collected.
Arm/Group | Haloperidol + Lorazepam | Loxapine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 120 minutes
Arm/Group | Haloperidol + Lorazepam | Loxapine
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/00/NCT03110900/Prot_SAP_000.pdf
  • Informed Consent Form (2017-09-26): https://cdn.clinicaltrials.gov/large-docs/00/NCT03110900/ICF_001.pdf